CLINICAL TRIAL: NCT03150238
Title: A Multicenter Prospective Cohort Study of Surgically Resected Crohn's Disease Patients Aiming to Identify Prognostic Factors for Re-operation: a New Score
Brief Title: Surgically Resected Crohn's Disease Patients: Prognostic Factors for Re-operation and New Score Building
Acronym: POCD2017
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Italian Group for the study of Inflammatory Bowel Disease (IG-IBD) (Other)
Responsible Party: Sponsor
Other Study IDs: 1687
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-operative Crohn Disease patients: Adult patients, with a defined diagnosis of CD, who underwent a surgery for CD in the previous 6 months
  Interventions: Other: observation of prognostic factors for relapse

INTERVENTIONS:
Other: observation of prognostic factors for relapse — The identification of the most relevant prognostic factors and the definition of their weight in predict the risk of re-intervention will be the basis for the definition of a combined score

SUMMARY:
The project will consist of a multicentre, prospective, observational study with a total duration of 24 months. Clinical, endoscopic and ultrasound data will be collected in a dedicated database (on IG-IBD Register), which will be used to identify potential clinical, endoscopic and ultrasound risk factors of re-operation. These data could be merged into a shared score, to stratify patients according to the risk of post-surgical re- operation and to define an optimal therapeutic management in the post- operative period. Approximately 220 adult patients, with a defined diagnosis of CD, who underwent a surgery for CD in the previous 6 months will be enrolled.

DETAILED DESCRIPTION:
Patients will be consecutively enrolled in this prospective cross-sectional study, during the first 12 months, and then followed for 12 (minimum) up to 24(maximum) months, depending on date of patients' enrolment (total study length: 2 years). Patients will be stratified according to risk factors and type of treatment carried out in that year

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 65 years, inclusive
* Diagnosis of Crohn's Disease (CD) for at least 6 months prior to enrolment, by clinical, endoscopic and histopathologic evidence
* First surgery for CD performed less than 6 months before enrolment (no second surgery allowed)
* Ability to provide written informed consent and to be compliant with the schedule of protocol assessments

Exclusion Criteria:

* Diagnosis of ulcerative colitis or indeterminate colitis
* Crohn's disease isolated at stomach, duodenum, jejunum, or perianal region, without ileo-colonic involvement
* More than one surgery for luminal CD
* Current stoma or need for ileostomy or colostomy
* Clinically relevant diseases making interpretation of the trial difficult or that would put the patient at risk of severe complications, in the opinion of the investigator
* Inability to provide written informed consent and poor compliance with the schedule of protocol assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, with a defined diagnosis of CD, who underwent a surgery for CD in the previous 6 months
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Re-operation rate in CD patients who underwent surgery for the first time - Re-operation rate | 12 months
  re-operation rate

SECONDARY OUTCOMES:
Ideation of a new score for the risk of re-operation in CD patients | 12 months
  The identification of the prognostic relevant factor and the evaluation of their specific weight in predicting the risk of re-intervention will be the basis for the ideation of a new score for the risk of re-operation in CD patients.

OTHER OUTCOMES:
Wall sonographic thickness | 12 months
  Wall sonographic thickness will be measured, to define, if feasible, a precise cut-off of thickness that could predict the risk of re-intervention, by a correlation with Rutgeerts' score

CONTACTS AND LOCATIONS:
Overall Officials: Federica Furfaro, MD, phD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
TO BE DETERMINED